CLINICAL TRIAL: NCT02779335
Title: Enteral Formula Tolerance in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15.09.US.HCN
Record Dates: First submitted 2016-03-18; First posted 2016-05-20 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-03

CONDITIONS: Enteral Nutrition
Keywords: tube-fed; Formula Tolerance; Pediatric Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enteral formula tube feeding (Other): Enteral fed children, ages 1-13, with establish enteral feeding access
  Interventions: Other: Enteral Formula

INTERVENTIONS:
Other: Enteral Formula — pediatric subjects will be fed a standard pediatric enteral formula tube feeding

SUMMARY:
The purpose of this prospective study seeks to assess ability to achieve enteral feeding goals with standard polymeric enteral formula in a stable, pediatric tube-fed population.

DETAILED DESCRIPTION:
In this prospective study, a population of stable, tube-fed children will consume a standard polymetric tube feeding formula to assess ability to achieve enteral feeding goals and tolerance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1 - 13 years of age
* Currently tolerating enteral feeding
* Has enteral access
* Requires enteral tube feeding to provide 90% or more of their nutritional needs (without the use of modular(s)) for at least 9 days
* Having obtained his/her and/or his/her legal representative's informed consent

Exclusion Criteria:

* Condition which contraindicates enteral feeding (i.e. intestinal obstruction)
* Lack of enteral access
* Any condition that would contraindicate use of the study product (i.e. need for severe fluid restriction, cow's milk protein allergy, other)
* Judged to be at risk for poor compliance to the study protocol
* Lack of informed consent
* Currently participating in another conflicting clinical trial

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Daily percentage of caloric nutritional goal met | 9 days

SECONDARY OUTCOMES:
Daily percentage of protein goal met | 9 days
Daily assessment of gastrointestinal tolerance - stool consistency | 9 days
  Daily assessment of stool consistency (liquid, formed, soft)
Daily assessment of gastrointestinal tolerance- Stool frequency | 9 days
  Daily assessment of number of stool
Daily assessment of gastrointestinal tolerance- Vomit | 9 days
  Daily assessment of frequency of vomit
Daily assessment of gastrointestinal tolerance - Flatulence | 9 days
  Daily assessment of presence of flatulence
Daily assessment of gastrointestinal tolerance - Abdominal pain | 9 days
  Daily assessment of abdominal pain
Frequency and nature of adverse events | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Minor, MMS, PA-C, Principal Investigator — Children's Center for GI and Nutrition
Locations (1):
- Children's Center for GI and Nutrition, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No